CLINICAL TRIAL: NCT02954250
Title: Modified Mindfulness Based Cognitive Therapy for the Treatment of Depressive Symptoms and Cognitive Inhibition in Patients at Risk for Suicide: A Pilot Randomized Controlled Trial
Brief Title: Mindfulness Based Cognitive Therapy for Depression and Cognitive Inhibition in Suicide
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Lady Davis Institute (Other)
Responsible Party: Principal Investigator, Dr. Karl Looper, Psychiatrist-in-Chief, Jewish General Hospital; Associate Professor, Dept. of Psychiatry, McGill University; Co-Lead, Geri-PARTy Research Group, Lady Davis Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IUSMD-16-17
Record Dates: First submitted 2016-09-20; First posted 2016-11-03 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Depression, Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Patients randomized to the control group will be offered literature on mental health promotion and Treatment as usual
- Mindfulness Group (Experimental): The intervention will consist of group, lasting 90 minutes in one session per week for 8 weeks. The exercises will be 5 minutes long alternating between 4 or 5 each session.
  Interventions: Behavioral: Mindfulness Based Cognitive Therapy

INTERVENTIONS:
Behavioral: Mindfulness Based Cognitive Therapy — The 8-week MMBCT protocol combines the practice of specific meditation techniques with cognitive therapy principles applicable to anxiety and depression. Each session will cover a meditation practice, as well as a relevant topic for discussion. The initial sessions will introduce general concepts of mindfulness (non-judgemental awareness, being in the moment, fostering curiosity, etc.), which will be expanded to more elaborate notions that are particularly relevant to anxiety, depression and suicidal ideations (recognizing thoughts are not facts, cultivating loving kindness for oneself, improving communication with others, etc.) Participants will be encouraged to practice the mindfulness techniques between sessions, a process that will be reviewed during groups in an ongoing fashion.
  Arms: Mindfulness Group

SUMMARY:
Background: According to the World Health Organization, one million people die by suicide each year worldwide and the rate of attempted suicide is ten times greater. A less known fact is that suicide is 3 times more frequent in elderly adults compared to younger counterpart. Unfortunately, predicting and preventing suicidal behaviours (SB) in general, and in elderly in particular, remain difficult. Clinical, biological and genetic data suggests that SB may be best understood according to a stress-vulnerability model where, more vulnerable individuals are at increased risk of committing a suicidal act when experiencing (mostly social) stress. Vulnerability to SB has also been associated with specific (i.e. distinct from comorbid psychiatric disorders like depression) neurocognitive alterations. However, the neurocognitive basis of suicidal behavior in elderly has been more rarely investigated.

Aim: Mindfulness based cognitive therapy (MBCT) has been successfully used to treat many psychiatric symptoms in many different populations, given that this therapy reduces cognitive creativity. Thus, this pilot study aims at addressing the SB in older adults with a Modified Mindfulness Based Cognitive Therapy (MMBCT).

Hypotheses: We hypothesise that MMBCT is not only a feasible intervention in older people with SB, but also, effective to treat depressive symptoms and suicidal ideation. Additionally, we will explore the changes in cognitive testing.

Methods: This is a pilot randomized controlled trial of a MMBCT tailored to older adults with depression and suicidal behaviors at the Douglas Mental Health University Institute. Patients with depression Hamilton Depression Rating Scale (HAM-D) >10 and suicidal ideation (Scale for Suicide Ideation [SSI] score ≥1) will be randomized to MMBCT or usual care. The meditation intervention will involve doing seated 90minute/week meditation exercises for 8 weeks. The primary outcomes will examine feasibility and acceptability of the treatment. The secondary outcome measures will scores in HAM-D and we will control for any important covariates differing between groups, (e.g. age, sex, # medical illnesses).

Perspectives: Implementation of these interventions could potentially prevent many consultations to psychiatry/mental health professionals. Increase quality of life, decrease medical comorbidity, illness and mortality. [2] Taken together, in our rapidly aging population, this could translate to substantial savings in health costs.

ELIGIBILITY:
Inclusion Criteria:

* Current major depressive episode, major depressive disorder (DSM-V) as per the HAM-D-21 ≥ 10;
* With no recent psychotropic modifications;
* History of suicidal ideation and/or personal history of suicide attempt;
* Normal cognition or Mild Cognitive Impairment ("Normal" Result on the 3-minute Mini-Cog Test).

Exclusion Criteria:

* Mild, Moderate, or Severe Dementia ("Abnormal" Result on the 3-minute Mini-Cog Test)[48]
* Acute psychotic symptoms
* Acute Suicidal intent (within 48-72 hours)
* Hearing impairment not improved with hearing aids and/or sound amplification
* Unable to engage in a group meditation for physical or practical reasons
* Ongoing Active Psychotherapy (e.g. a course of CBT psychotherapy)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Fulfillment of initial recruitment goals (first 20 patients) | within 12 months

SECONDARY OUTCOMES:
Decreases in HAM-D Scale | over 8-weeks period
Improvement in the Stroop task performances | over 8-weeks period

CONTACTS AND LOCATIONS:
Locations (1):
- Douglas Mental Health University Institute, Montreal, Quebec, Canada